CLINICAL TRIAL: NCT01122966
Title: The Effect of Intracameral and Subconjunctival Injections of Bevacizumab in Trabeculectomy With Antimetabolite
Brief Title: The Effect of Bevacizumab on the Trabeculectomy
Acronym: bevazicumab
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Changwon Kee, Samsung Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-01-033
Record Dates: First submitted 2010-04-15; First posted 2010-05-13 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Glaucoma
Keywords: trabeculectomy
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- trabeculectomy (Other): Subjects who have trabeculectomies with intraocular bevacizumab injection
  Interventions: Drug: intraocular injections of bevacizumab

INTERVENTIONS:
Drug: intraocular injections of bevacizumab — intracameral and subconjunctival injections
  Other Names: glaucoma filtering surgery

SUMMARY:
The investigators plan to evaluate the additive effect of intracameral and subconjunctival injections of bevacizumab in trabeculectomies with other antimetabolites.

DETAILED DESCRIPTION:
Glaucoma filtration surgery is routinely utilized to control intraocular pressure in glaucomatous patients. It reduces IOP by creating a fistula between the anterior chamber and the subconjunctival space with a filtering bleb. Increased wound healing response affects the function and morphology of the filtering bleb, and wound healing involves a series of biological events beginning with hemostasis.

Corticosteroids and antifibrosis agents such as mitomycin C and 5-fluorouracil have been employed in trabeculectomy to delay wound healing and hence to improve the success rate of surgery by inhibiting inflammation and fibroblastic activity, and the use of these antiscarring agents is generally believed to improve the success rate of trabeculectomy.But this rate decreased with passing time and thus was not perfect.

Vascular endothelial growth factor is a pivotal stimulator of angiogenesis because its binding to VEGF receptors has been demonstrated to promote endothelial cell migration and proliferation in wound healing.Therefore, anti-VEGF agents may potentially modulate wound healing following glaucoma filtration surgery.

The principal objective of this study was to evaluate the additive effect of intracameral and subconjunctival injections of bevacizumab in trabeculectomy.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma patients who have trabeculectomy

Exclusion Criteria:

* patients with the other ocular disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure | on postoperative 1month
  Intraocular pressure is planned to measure when the patient visit the clinic. All intraocular pressure measurements is acquired by glaucoma specialists, using a slitlamp-mounted Goldmann applanation tonometer.

SECONDARY OUTCOMES:
intraocular pressure | on postoperative 6months, 12months, 18months, 24months
  Intraocular pressure is planned to measure when the patient visit the clinic. All intraocular pressure measurements is acquired by glaucoma specialists, using a slitlamp-mounted Goldmann applanation tonometer.

CONTACTS AND LOCATIONS:
Overall Officials: Changwon Kee, M.D., Ph.D, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Li Z, Van Bergen T, Van de Veire S, Van de Vel I, Moreau H, Dewerchin M, Maudgal PC, Zeyen T, Spileers W, Moons L, Stalmans I. Inhibition of vascular endothelial growth factor reduces scar formation after glaucoma filtration surgery. Invest Ophthalmol Vis Sci. 2009 Nov;50(11):5217-25. doi: 10.1167/iovs.08-2662. Epub 2009 May 27. PMID 19474408
- [Background] Grewal DS, Jain R, Kumar H, Grewal SP. Evaluation of subconjunctival bevacizumab as an adjunct to trabeculectomy a pilot study. Ophthalmology. 2008 Dec;115(12):2141-2145.e2. doi: 10.1016/j.ophtha.2008.06.009. Epub 2008 Aug 9. PMID 18692246